CLINICAL TRIAL: NCT02438111
Title: The Role of the Gut Metagenome on the Development of Age Related Macular Degeneration (AMD)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: KEK BE 205/13, PB_2016-01922
Record Dates: First submitted 2015-04-28; First posted 2015-05-08 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Metagenome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood serum/ stool
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- age related macular degeneration: metagenome AMD
  Interventions: Genetic: metagenome
- controls: metagenome controls
  Interventions: Genetic: metagenome

INTERVENTIONS:
Genetic: metagenome — metagenome

SUMMARY:
The primary objective of this study is to assess whether compositional and functional alterations of the gut metagenome may be related to AMD. The primary variable for this assessment is the composition of the gut metagenome which will be analyzed by shotgun sequencing to characterize the faecal metagenome. The secondary endpoint is to assess whether single nucleotide polymorphisms in CFH, ARMS2, C3, PLEKHA1, HTRA-1, VEGF-A, VEGF-B, VEGFR and APOE genes which have been shown to be risk factors for the development of AMD and other macular diseases correlate with alterations in the gut metagenome .

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is the most frequent cause of blindness in the elderly. Despite major research efforts in the last decades the etiology of AMD remains largely undefined and therefore treatment options are only very limited. However, there is evidence that nutrition and inflammation play a role in the pathogenesis of AMD . The latter is also corroborated by the finding that single nucleotide polymorphism in the gene encoding complement factor H is associated with AMD . In addition to CHF other genes such as ARMS2, C3, PLEKHA1, HTRA-1, VEGF-A, VEGF-B, VEGFR and APOE have been associated with development of AMD. Recent findings have implicated the gut microbiota as a contributor of metabolic diseases through the modulation of host metabolism and inflammation . Gut bacteria use mostly fermentation to generate energy, converting sugars, in part, to short-chain fatty acid, that are used by the host as energy source. Beyond short-chain fatty acids gut bacteria can provide some amino acids and contribute certain vitamins such as biotin to the host . The investigators propose to investigate whether compositional and functional alterations of the gut microbiota are a risk factor for developing AMD.

ELIGIBILITY:
Inclusion criteria:

* Subject must be willing to give written informed consent and willing to provide blood and stool probes
* Patients with clinically confirmed AMD 18 years of age or greater
* Probands with no signs of AMD 18 years of age or greater

Exclusion criteria:

* Smoking
* Chronic inflammatory disease (autoimmune diseases such as rheumatoid arthritis, lupus erythematodes, chronic inflammatory bowel disease)
* Diabetes as defined by The World Health Organization (WHO) criteria
* Treated hyperlipidemia
* Obesity with a body mass index (BMI) greater than or equal to 30
* Recent (3 month) history of use of systemic antibiotics
* Opacities of ocular media excluding detailed observation of the retina

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with age related macular degeneration (AMD)
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2013-12; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
taxonomic and functional characterization of gut microbiota | 3 years

SECONDARY OUTCOMES:
Gut-microbiota-based AMD classification | 3 years
AMD-associated gut microbial markers | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Martin Zinkernagel, M.D, PhD, Study Chair — Department of Ophthalmology, University Hospital Bern, Switzerland; Martin S Zinkernagel, MD, PhD, Principal Investigator — Department of Ophthalmology, University Hospital Bern, Switzerland; Martin Fiedler, MD, Study Director — University Hospital Bern, Switzerland
Locations (1):
- Inselspital Bern, Department of Ophthalmology, Bern, Switzerland

REFERENCES:
- [Derived] Sporri L, Studer JM, Kreuzer M, Rotzetter J, Scharer D, Largiader CR, Jaggi D, Zinkernagel MS, Zysset-Burri DC. Linking the microbiome to the complement system in geographic atrophy. NPJ Genom Med. 2026 Feb 2. doi: 10.1038/s41525-026-00550-7. Online ahead of print. PMID 41629364